CLINICAL TRIAL: NCT03775954
Title: Fetal Electrophysiologic Abnormalities in High-risk Pregnancies Associated With Fetal Demise
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Wisconsin, Madison (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Shared Medical Technology, Inc. (Industry); Tristan Technologies, Inc (Unknown)
Responsible Party: Principal Investigator, Janette F. Strasburger, Professor, Medical College of Wisconsin
Other Study IDs: PRO00031598; R01HL143485 (NIH)
Record Dates: First submitted 2018-10-24; First posted 2018-12-14 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: High Risk Pregnancy; Congenital Heart Disease; Fetal Hydrops; Twin Monochorionic Monoamniotic Placenta; Gastroschisis; Fetal Demise; Stillbirth; Fetal Arrhythmia; Long QT Syndrome; Intrauterine Fetal Death; Sudden Infant Death; Pregnancy Loss; Twin Twin Transfusion Syndrome; Birth Defect; Fetal Cardiac Anomaly; Fetal Cardiac Disorder; Fetal Death; Brugada Syndrome
Keywords: Fetal Magnetocardiography; Stillbirth; Intrauterine Fetal Demise; Mobile Medical Technologies; Fetal Heart Rate Variability; Fetal Arrhythmias; High Risk Pregnancy; Pregnancy; Fetal Anomaly; Fetal Echocardiography; Non-Stress Testing; New Technology; Birth Defects; Fetal Research
MeSH Terms: conditions — Heart Defects, Congenital; Hydrops Fetalis; Gastroschisis; Fetal Death; Stillbirth; Long QT Syndrome; Sudden Infant Death; Fetofetal Transfusion; Congenital Abnormalities; Brugada Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1) Fetal Congenital Heart Disease: Pregnancy with major fetal congenital heart disease, after 20 weeks gestation, and as neonate following delivery. Two fetal magnetocardiograms (fMCG) and 1 neonatal electrocardiogram (nECG) will be obtained and heart rate, rhythm, and conduction patterns will be compared.
  Interventions: Diagnostic Test: Fetal Magnetocardiogram and Neonatal Electrocardiogram
- 2) History of fetal demise (Stillbirth): Pregnancy with a history of an unexplained fetal demise (stillbirth at 20 -40 weeks gestation) during any prior pregnancy. Two fetal magnetocardiograms (fMCG) and 1 neonatal electrocardiogram (nECG) will be obtained and heart rate, rhythm, and conduction patterns will be compared.
  Interventions: Diagnostic Test: Fetal Magnetocardiogram and Neonatal Electrocardiogram
- 3) Fetal hydrops, immune or non-immune: Pregnancy with fetal hydrops, immune or non-immune, at or after 20 weeks gestation. Two fetal magnetocardiograms (fMCG) and 1 neonatal electrocardiogram (nECG) will be obtained and heart rate, rhythm, and conduction patterns will be compared.
  Interventions: Diagnostic Test: Fetal Magnetocardiogram and Neonatal Electrocardiogram
- 4) Fetal gastroschisis: Pregnancy with fetal gastroschisis, at or after 20 weeks gestation. Two fetal magnetocardiograms (fMCG) and 1 neonatal electrocardiogram (nECG) will be obtained and heart rate, rhythm, and conduction patterns will be compared.
  Interventions: Diagnostic Test: Fetal Magnetocardiogram and Neonatal Electrocardiogram
- 5) Twin pregnancy, monochorionic: Twin pregnancy, monochorionic, with or without twin-twin transfusion syndrome, at or after 20 weeks gestation. Two fetal magnetocardiograms (fMCG) and 1 neonatal electrocardiogram (fMCG) will be obtained and heart rate, rhythm, and conduction patterns will be compared.
  Interventions: Diagnostic Test: Fetal Magnetocardiogram and Neonatal Electrocardiogram

INTERVENTIONS:
Diagnostic Test: Fetal Magnetocardiogram and Neonatal Electrocardiogram — Fetal Magnetocardiography (fMCG) is a new non-invasive diagnostic procedure that records tiny fetal cardiac signals similar to an Electrocardiogram or Holter monitor. The magnetometer has FDA clearance, and does not emit magnetic, electric or other energies. This is not an MRI. Examples of fetal MCG's can be found in the Links. The American Heart Association Scientific Statement on Fetal Diagnosis and Treatment (Circulation, 2014) has declared fMCG to be Class IIa for fetal heart rhythm abnormalities, meaning that benefit far exceeds risk. As part of this study, a neonatal electrocardiogram (nECG) will be obtained for comparison after the baby is born.

SUMMARY:
Each year world-wide, 2.5 million fetuses die unexpectedly in the last half of pregnancy, 25,000 in the United States, making fetal demise ten-times more common than Sudden Infant Death Syndrome. This study will apply a novel type of non-invasive monitoring, called fetal magnetocardiography (fMCG) used thus far to successfully evaluate fetal arrhythmias, in order to discover potential hidden electrophysiologic abnormalities that could lead to fetal demise in five high-risk pregnancy conditions associated with fetal demise.

DETAILED DESCRIPTION:
Fetal demise occurs in over 25,000 pregnancies annually in the US and over 2.5 million in pregnancies worldwide. Certain maternal-fetal-placental abnormalities can have a high risk of fetal demise. Despite advances in fetal surveillance with ultrasound and cardiotocography, the reduction in fetal mortality lags behind that of the neonate and has shown little decline in the past decade. This suggests that the type of fetal monitoring used may not be assessing the correct indicators of mortality. In all other age groups, electrocardiographic (ECG) and continuous heart rate (HR) monitoring are used in every intensive care unit or emergency setting; however, for the fetus, the ECG signal is nearly completely insulated and inaccessible. As the result, indirect assessment of cardiac rhythm is obtained using echocardiography/Doppler, but echo/Doppler does not have the precision to assess beat-to-beat HR variability and cannot assess cardiac repolarization at all. In this study, the investigators will evaluate five high risk conditions (major congenital heart disease in the fetus, fetal hydrops (immune and non-immune), monochorionic twin pregnancy, prior pregnancy ending in fetal demise, and gastroschisis) using Fetal Magnetocardiography (fMCG)which detects the natural magnetic signals accompanying the cardiac electrical signal. It is a new, safe, and non-invasive recording technique that has been performed for several decades, and has recently gained FDA approval for recording cardiac signals at all ages, including in the fetus. Normative data has been obtained at the University of Wisconsin - Madison Biomagnetism Laboratory in 257 healthy fetuses by co-investigator Ronald T. Wakai, PhD. Over 550 serious fetal arrhythmias have been evaluated to date. Fetal MCG has proven invaluable in fetal Long QT Syndrome in identifying markers for risk of sudden death such as Torsades de Pointes Ventricular Tachycardia (VT), T wave alternans, 2nd degree AV block, and QTc>590 ms. To date, fMCG has not been systematically applied to diseases that are not associated with recognizable arrhythmias because the impact of silent conduction and repolarization defects has been underappreciated. In this grant, the investigators hypothesize that beat-to-beat fetal heart rate variability abnormalities and electrophysiologic abnormalities, are present in five high risk maternal-fetal-placental conditions associated with fetal demise. The study will determine which electrophysiologic abnormalities precede fetal demise or adverse pregnancy outcome. Preliminary findings in healthy normal subjects in RO1HL063174 (Wakai) show repolarization abnormalities in up to 5%, and some of these are modifiable once recognized. Two hundred pregnant subjects will be studied over a 5 year period both at referral (~20-27 weeks GA) and later in pregnancy at 30-37 weeks GA. fMCG results will be compared to neonatal ECG (nECG) obtained at 0-4 weeks of life. This will determine whether specific abnormal heart rate, rhythm and conduction patterns emerge that characterize the condition, which will then allow the high risk obstetrician to better predict risk of fetal demise in the future.

ELIGIBILITY:
Inclusion Criteria:

* Current pregnancy complicated by one of the five diagnostic categories

  * prior unexplained Stillbirth at/after 20 weeks gestation
  * fetal major congenital heart defect
  * fetal hydrops
  * fetal gastroschisis
  * monochorionic twin pregnancy
* Subject must be 18 years of age or older
* Subject must be English speaking and must be able to read and sign the consent form in English
* Subject must be able to recline comfortably for 1-3 hours
* Subject must be willing to complete all three procedures (fMCG, fMCG, nECG) as per protocol, unless medically unable
* Subject must be willing to allow us to review her and her infants prenatal, deliver, and post-natal records to verify diagnosis, and clinical findings.

Exclusion Criteria:

* Severe claustrophobia not reduced by taking breaks, or by having the light on, or by having someone in the room with them.
* Active labor
* Acute illness
* Unable to recline comfortably with a pillow for more than 1-3 hours (assuming some breaks are provided)
* Weight over 450 lbs
* An electric stimulation device (TENS unit, pacemaker, or nerve stimulator) that could produce electric or magnetic noise.

  * Note that the Tristan 624 Magnetometer does not pose a risk to the subject's device, (since fMCG does not produce any energy or magnetism), but stimulators themselves can cause interference for our recordings. Some devices may still qualify, and discussion with study nurse may be useful if subject has a pacemaker or similar device.

The subject will have a single 2-3 hour fetal magnetocardiogram at approximately 20 and 27 weeks GA, and again, if medical condition allows, between 30 and 37 weeks GA, then her infant will have an ECG between 0 and 4 weeks of age. Subjects will be paid a nominal fee for their participation each time, as well as transportation reimbursement if >25 miles. For subjects traveling a long distance, the ECG may be performed locally or at home.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study involves pregnant women and subsequently-born neonate(s) of either gender.
Study Population: Current pregnancy complicated by one of the five diagnostic categories (fetal major congenital heart disease, prior unexplained Stillbirth at/after 20 weeks gestation, fetal hydrops, fetal gastroschesis, or monochorionic twin pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability using fMCG | Comparison of procedures at approximately 20-27 weeks gestation, at 30-37 weeks gestation, and at neonatal ECG at 0-4 weeks of age
  To measure and compare the fMCG heart rate variability in five pregnancy conditions associated with fetal demise, to those of gestation matched normal fetuses.
Cardiac conduction | Comparison of cardiac time intervals at approximately 20-27 weeks gestation, 30-37 weeks gestation and at neonatal ECG at 0-4 weeks of age
  To measure and compare the fMCG cardiac time intervals in five pregnancy conditions associated with fetal demise, to those of gestation matched normal fetuses and to neonatal ECGs at 0-4 weeks of age.
Cardiac repolarization | Comparison of cardiac repolarization at approximately 20-27 weeks gestation, 30-37 weeks gestation and neonatal ECG at 0-4 weeks of age.
  To measure and compare the fMCG cardiac repolarization patterns in five pregnancy conditions associated with fetal demise, to those of gestation matched normal fetuses, and to neonatal ECGs at 0-4 weeks of age.

SECONDARY OUTCOMES:
Unique "signature" electrophysiologic abnormalities | Comparison of findings at approximately 20-27 weeks gestation, 30-37 weeks gestation and neonatal ECG at 0-4 weeks of age
  2a) To determine whether unique "signature" electrophysiologic abnormalities are present in any of these five maternal-fetal diseases, and 2b) to define at what trimester these develop. Understanding any unique findings could allow study of specific treatment strategies in the future.
  findings are first seen.
Pregnancy outcomes | Comparison of findings at approximately 20-27 weeks gestation, 30-37 weeks gestation and neonatal ECG at 0-4 weeks of age
  To correlate fMCG findings with 3a) outcomes of pregnancies (fetal demise, premature delivery, small for GA, 5 minute APGAR < 5, neonatal death) and 3b) fMCG cardiac time intervals with postnatal ECG intervals at 0-4 weeks of age.

CONTACTS AND LOCATIONS:
Overall Officials: Janette F Strasburger, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Only de-identified data can be released

REFERENCES:
- [Background] Donofrio MT, Moon-Grady AJ, Hornberger LK, Copel JA, Sklansky MS, Abuhamad A, Cuneo BF, Huhta JC, Jonas RA, Krishnan A, Lacey S, Lee W, Michelfelder EC Sr, Rempel GR, Silverman NH, Spray TL, Strasburger JF, Tworetzky W, Rychik J; American Heart Association Adults With Congenital Heart Disease Joint Committee of the Council on Cardiovascular Disease in the Young and Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and Council on Cardiovascular and Stroke Nursing. Diagnosis and treatment of fetal cardiac disease: a scientific statement from the American Heart Association. Circulation. 2014 May 27;129(21):2183-242. doi: 10.1161/01.cir.0000437597.44550.5d. Epub 2014 Apr 24. PMID 24763516
- [Background] Strasburger JF, Wakai RT. Fetal cardiac arrhythmia detection and in utero therapy. Nat Rev Cardiol. 2010 May;7(5):277-90. doi: 10.1038/nrcardio.2010.32. PMID 20418904
- [Background] Cuneo BF, Strasburger JF, Yu S, Horigome H, Hosono T, Kandori A, Wakai RT. In utero diagnosis of long QT syndrome by magnetocardiography. Circulation. 2013 Nov 12;128(20):2183-91. doi: 10.1161/CIRCULATIONAHA.113.004840. PMID 24218437
- [Background] Batie M, Bitant S, Strasburger JF, Shah V, Alem O, Wakai RT. Detection of Fetal Arrhythmia Using Optically-Pumped Magnetometers. JACC Clin Electrophysiol. 2018 Feb;4(2):284-287. doi: 10.1016/j.jacep.2017.08.009. No abstract available. PMID 29527577
- [Background] Strand S, Strasburger JF, Cuneo BF, Wakai RT. Complex and Novel Arrhythmias Precede Stillbirth in Fetuses With De Novo Long QT Syndrome. Circ Arrhythm Electrophysiol. 2020 May;13(5):e008082. doi: 10.1161/CIRCEP.119.008082. Epub 2020 May 18. PMID 32421437
- [Background] Strand S, Lutter W, Strasburger JF, Shah V, Baffa O, Wakai RT. Low-Cost Fetal Magnetocardiography: A Comparison of Superconducting Quantum Interference Device and Optically Pumped Magnetometers. J Am Heart Assoc. 2019 Aug 20;8(16):e013436. doi: 10.1161/JAHA.119.013436. Epub 2019 Aug 9. PMID 31394997
- [Background] Wacker-Gussmann A, Strasburger JF, Wakai RT. Fetal Magnetocardiography Alters Diagnosis and Management in Fetal Congenital Heart Disease and Cardiomyopathy. JACC Clin Electrophysiol. 2022 Sep;8(9):1159-1161. doi: 10.1016/j.jacep.2022.04.012. Epub 2022 Jun 29. No abstract available. PMID 36137723
- [Background] Wacker-Gussmann A, Strasburger JF, Wakai RT. Contribution of Fetal Magnetocardiography to Diagnosis, Risk Assessment, and Treatment of Fetal Arrhythmia. J Am Heart Assoc. 2022 Aug 2;11(15):e025224. doi: 10.1161/JAHA.121.025224. Epub 2022 Jul 29. PMID 35904205
- [Background] Strasburger JF, Eckstein G, Butler M, Noffke P, Wacker-Gussmann A. Fetal Arrhythmia Diagnosis and Pharmacologic Management. J Clin Pharmacol. 2022 Sep;62 Suppl 1(Suppl 1):S53-S66. doi: 10.1002/jcph.2129. PMID 36106782
- See also: Fetal MCG Research — https://www.medphysics.wisc.edu/wp/research/biomagnetism/
- See also: Children's Hospital of Wisconsin Herma Heart Institute — https://childrenswi.org/medical-care/herma-heart
- See also: NIH Seminar Dr. Strasburger is co-chair, speaks at 32 minutes, Dr. Wakai speaks at 62 minutes on fMCG and a participant speaks at 1::37 minutes on her experience in our study. — https://datascience.nih.gov/news/nih-virtual-workshop-near-term-applications-of-quantum-sensing-technologies-in-biomedical-sciences